CLINICAL TRIAL: NCT02820610
Title: Dexmedetomidine Versus Magnesium Sulfate as an Adjuvant to Intraperitoneal Bupivacaine for Pain Relief in Children Undergoing Laparoscopic Herniorrhaphy: a Randomized Controlled Study.
Brief Title: Intraperitoneal Analgesia in Pediatric Laparoscopy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Seham Mohamed Moeen Ibrahim, lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SM62016
Record Dates: First submitted 2016-06-29; First posted 2016-07-01 (Estimated); Last update posted 2020-01-03 (Actual); Status verified 2020-01

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia | interventions — Dexmedetomidine; Magnesium Sulfate; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dexmedetomidine (Active Comparator): 2 mg/kg bupivacaine 0.5% and 1 ug/kg of dexamedetomidine diluted in normal saline 0.9 % will instilled into the peritoneal cavity
  Interventions: Drug: Dexmedetomidine
- Magnesium sulfate (Active Comparator): 2 mg/kg bupivacaine 0.5% and 30 mg/kg of magnesium sulfate diluted in normal saline 0.9 % will instilled into the peritoneal cavity
  Interventions: Drug: Magnesium Sulfate
- Control group (Placebo Comparator): 2 mg/kg bupivacaine 0.5% diluted in normal saline 0.9 % will instilled into the peritoneal cavity.
  Interventions: Drug: Normal saline 0.9 %

INTERVENTIONS:
Drug: Dexmedetomidine — 2 mg/kg bupivacaine 0.5% and 1 ug/kg of dexamedetomidine diluted in normal saline 0.9 % will instilled into the peritoneal cavity
  Other Names: Presidx
  Arms: Dexmedetomidine
Drug: Magnesium Sulfate — 2 mg/kg bupivacaine 0.5% and 30 mg/kg of magnesium sulfate diluted in normal saline 0.9 % will instilled into the peritoneal cavity
  Arms: Magnesium sulfate
Drug: Normal saline 0.9 % — 2 mg/kg bupivacaine 0.5% diluted in normal saline 0.9 % will instilled into the peritoneal cavity.
  Arms: Control group

SUMMARY:
It is important to keep children undergoing laparoscopic surgery pain free with rapid return to normal activity.

DETAILED DESCRIPTION:
Pain following laparoscopy is less intense than after laparotomy. Nevertheless, laparoscopy is not pain free and control of post-laparoscopy pain remains a major concern. The exact cause of such pain remains uncertain, and yet, diaphragmatic irritation and peritoneal stretching associated with gas insufflation may be responsible for shoulder and diffuse abdominal pain.

additionally poor pain control could limit the activity of children following laparoscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

1. age (1 to 6 years)
2. ASA physical status I or II.
3. scheduled for laparoscopic hernia repair under general anesthesia.

Exclusion Criteria:

1. Allergy to study drugs,
2. Receiving chronic pain treatment, antiepileptic therapy or magnesium therapy,
3. sever hepatic or renal impairment,

Ages: 1 Year to 6 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 97 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Postoperative pain | 48 hr
  The Face Legs Activity Cry and Consolability (FLACC) pain score

SECONDARY OUTCOMES:
the functional recovery | 48 hours after surgery
  the functional activity score (FAS)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Assuit University, Asyut, Assuit, Egypt

IPD SHARING:
Plan to Share IPD: Yes